CLINICAL TRIAL: NCT04964752
Title: Effectiveness and Safety Study of the Continuous Glucose Monitoring System for Home Use (Including In-clinic Sessions) in Patients With Diabetes
Brief Title: A Study of the Continuous Glucose Monitoring System for Home Use in Patients With Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: Powder (Guangzhou) Pharmaceuticals Limited (Unknown); Powder Pharmaceuticals (HK) Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PL-CGM-202006
Record Dates: First submitted 2021-07-11; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- the upper arm group on Day 2 (Other): The upper arm group to perform Visit 3 venous blood glucose measurement on Day 2.
  Interventions: Device: continuous glucose-monitoring
- the upper arm group on Day 15±1 day (Other): The upper arm group to perform Visit 3 venous blood glucose measurement on Day 15±1 day.
  Interventions: Device: continuous glucose-monitoring
- the upper arm group on Day 29±1 day (Other): The upper arm group to perform Visit 3 venous blood glucose measurement on Day 29±1 day.
  Interventions: Device: continuous glucose-monitoring
- the abdomen group on Day 2 (Other): The abdomen group to perform Visit 3 venous blood glucose measurement on Day 2.
  Interventions: Device: continuous glucose-monitoring
- the abdomen group on Day 15±1 (Other): The abdomen group to perform Visit 3 venous blood glucose measurement on Day 15±1.
  Interventions: Device: continuous glucose-monitoring
- the abdomen group on Day 29±1 (Other): The abdomen group to perform Visit 3 venous blood glucose measurement on Day 29±1.
  Interventions: Device: continuous glucose-monitoring

INTERVENTIONS:
Device: continuous glucose-monitoring — Continuous glucose-monitoring device indicated for continually recording interstitial fluid glucose levels in patients with diabetes.
  Other Names: CGM

SUMMARY:
Subjects in the upper arm group will have a sensor of the CGM System inserted on each arm (left and right upper arm). Subjects in the abdomen group will have 2 sensors inserted, one on each side of the abdomen (left and right abdomen) The sensors will be placed for 29 days. After sensor insertion, the CGM system should be calibrated with capillary blood glucose readings from a self-monitoring blood glucose meter。

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or 2 diabetes mellitus
2. Male or female age ≥ 18 years old and ≤ 70 years old
3. Willingness to adopt measures to prevent water coming into contact with the device sensor (e.g. abstain from swimming, sauna, avoid hitting the sensor with direct jets of water)
4. Ability to communicate with the investigators, able to operate medical device after training and comply with the testing procedures outlined in this protocol (including, but not limited to, willing to wear the continuous glucose monitor and testing capillary blood glucose)
5. Subjects who show understanding of the study procedures and willing to sign a written informed consent form.

Exclusion Criteria:

1. Hospitalization due to diabetic ketoacidosis or severe hypoglycemia, within 3 months prior to screening
2. HbA1c >13% or urine ketone 3+
3. Use of pacemaker
4. Body Mass Index (BMI) ≤18.0kg/m2
5. Extensive skin changes/diseases that preclude wearing the required number of devices on normal skin at the proposed application sites, i.e. upper arm or abdomen (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis)
6. Any psychiatric disease such as depression or anxiety
7. Any severe hepatic, renal, cardiac, cerebral, respiratory or neurological diseases (e.g. serum ALT, AST, Creatinine level ≥3 times the upper limit of normal)
8. Has a MRI scan, CT scan or other procedure requiring the subject be under strong magnetic or electromagnetic environment, scheduled during the proposed study participation
9. Blood loss >400ml in the past 3 months (including blood donation)
10. Have a known allergy to medical-grade adhesives, or known hypersensitivity to any of the products used in the study
11. Difficulty in sampling venous blood or cannot tolerate venipuncture
12. Participated in other investigational studies in the past 3 months
13. Currently pregnant or lactating women, or positive pregnancy test
14. Any condition that, in the opinion of the investigator, renders the subject not suitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
%20/20 agreement between the test device readings and the EKF readings: %20/20 = A + B | up to 29 days
  A = the proportion of the CGM system values that were within ±20% of paired EKF values >4.4mmol/L (>80 mg/dL) B = the proportion of the CGM system values that were within ±1.1mmol/L (20mg/dL) of paired EKF values ≤4.4mmol/L (≤80mg/dL)
Proportion of readings in Region A + Region B of Clarke Error Grid | up to 29 days
  Analyze the proportion of readings in each region (Region A, B, C D and E). Readings in Region A are clinically accurate, while readings in Region B are of clinically acceptable accuracy. Readings in C, D and E are inaccurate to various degrees.
Proportion of readings in Region A + Region B of Consensus Error Grid | up to 29 days
  Analyze the proportion of readings in Region A and Region B.
the percentage of MARD (Mean Absolute Relative Difference) | up to 29 days
  Analyze the proportion of readings in MARD <18% (95%CI<20%).

SECONDARY OUTCOMES:
Alarm success rate1 | up to 29 days
  Hypoglycemia alarm success rate and failure rate (sensitivity)
Alarm success rate2 | up to 29 days
  Hypoglycemia detection rate and missed detection rate (specificity)
Alarm success rate 3 | up to 29 days
  Hyperglycemia alarm success rate and failure rate
Alarm success rate 4 | up to 29 days
  Hyperglycemia detection rate and missed detection rate
Sensor Stability | up to 29 days
  Compare the accuracy of the sensor between Day 2(22h~48h after insertion), Day 15±1day, Day 29±1day to evaluate sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chow, Prof., Principal Investigator — Prince of Wales Hospital, the Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No